CLINICAL TRIAL: NCT01329887
Title: Evaluation of the Effect of Ketanserine on Sublingual Microcirculation by SDF Imaging in Septic Patients on the Intensive Care
Brief Title: The Effect of Ketanserin on the Microcirculation in Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Dr, Frisius Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPO 736
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: microcirculation; SDF; ketanserin; severe sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ketanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- administration of ketanserin (Other)
  Interventions: Drug: ketanserin

INTERVENTIONS:
Drug: ketanserin — ketanserin administration is started and increase, guided by the effect on sublingual MFI, dosage is 0,03mg/kg/hr

SUMMARY:
This study is an evaluation of the effect of ketanserine on sublingual microcirculation in intensive care patients with severe sepsis.

DETAILED DESCRIPTION:
This is a pilot study, including 10 ICU patients with severe sepsis with MFI < 2,5 after fulfillment of a strict resuscitation protocol. At the start of the study, a baseline SDF measurement is made, when MFI < 2,5 inclusion in the study is permitted and intravenous ketanserin administration is started and subsequently increased, guided by the effect on sublingual MFI, until a safe maximum dosage is reached. Safety margins for hypotension are defined in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis and MFI < 2,5 after resuscitation

Exclusion Criteria:

* age < 18 year old
* pregnant
* participation other trials prolonged Qt interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
microcirculation | 2 hours
  achievement of a microvascular flow index >2,9

SECONDARY OUTCOMES:
ketanserine dosage | 48 hours
  obtaining a global indication of the ketanserin dosage needed to achieve a MFI >2,9 and the incidence of hypotension

CONTACTS AND LOCATIONS:
Overall Officials: E Boerma, MDPhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands